CLINICAL TRIAL: NCT05853614
Title: A Nurse-Led Intervention to Enhance Quality of Life Among Early Phase Clinical Trial Participants: A Pilot Study
Brief Title: Nurse-Led Quality of Life Study-Phase I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Oncology Nursing Society (Other)
Responsible Party: Principal Investigator, Debra Marie Lundquist, R.N., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-695
Record Dates: First submitted 2023-04-13; First posted 2023-05-11 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Quality of Life
Keywords: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurse-Led Quality of Life Intervention (Experimental): Participants and caregivers will complete study procedures as outlined:
  * Completion of surveys at four timepoints (baseline, one month, two months, and three months)
  * Three visits on-site with trained clinical research nursing staff.
  * Semi-structured exit interviews with participants and caregivers.
  Interventions: Behavioral: Quality of Life Intervention

INTERVENTIONS:
Behavioral: Quality of Life Intervention — Comprised of three components: (1) establishment of clinical research nurse (CRN) and patient relationship, (2) assessment and monitoring of physical, psychological, social, and spiritual well-being and patient-reported outcomes, and (3) weekly, interdisciplinary team meetings led by CRN.

SUMMARY:
The purpose of this study is to pilot test a brief, population-specific nurse-led, quality of life (QOL) intervention with early phase cancer clinical trial (EP-CT) participants.

The name of the intervention used in this research study is:

-Nurse-Led Quality of Life Intervention (comprised of nurse-patient relationship, assessment and monitoring of participant QOL, and interdisciplinary team meetings led by the CRN (clinical research nurse).

DETAILED DESCRIPTION:
This is a single-site study evaluating the feasibility and acceptability as well as patient-reported and clinical outcomes of a nurse-led, quality of life intervention with EP-CT participants.

The research study procedures include obtaining consent to participate, meeting with research nurses monthly for three months, completing questionnaires, and an interview with the study staff at the end of the study.

Participation in this research study is expected to be for a total of six months.

It is expected that about 35 people, 25 caregivers, and 10 clinicians will take part in this research study.

The Oncology Nursing Foundation is supporting this research study by providing funding.

ELIGIBILITY:
Patient Inclusion Criteria:

-> 18 years of age.

* Adults with cancer enrolled on an EP-CT in the Termeer Center at Massachusetts General Hospital.
* Able to read and respond to questions in English.

Caregiver Inclusion Criteria:

* A relative or friend of the eligible patient whom the patient identifies as being involved in their medical care.

  -> 18 years of age.
* Verbally fluent in English.

Clinician Inclusion Criteria:

* Clinician must be an oncology nurse.
* CRN for a minimum of 18 months.
* fulltime employee in the Termeer Center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Rate of Participant Enrollment | At screening
  The study will be feasible if at least 60% (95% confidence interval of +/-12%) enrollment of approached and eligible patients agree to participate in the study and sign informed consent
Rate of Participant Assessment Completion | Baseline to 3 months
  This study will be feasible if at least 70% (95% confidence interval of +/- 15%) of enrolled participants will complete a minimum of 60% of their patient-reported symptom assessments within the study period.
Intervention Acceptability | Baseline to 3 months
  Acceptability is defined as > 70% of patients, caregivers, and clinicians report favorable responses to the acceptability questions.

SECONDARY OUTCOMES:
Change in Quality of Life (QOL) | Baseline to 3 months
  Assessed by Functional Assessment of Cancer Therapy-General (FACT-G), a questionnaire comprised of 27 items with scale ratings validated to measure physical, emotional, social, and functional well-being of clinical trial participants.
Change in Symptom Burden | Baseline to 3 months
  Assessed through the Edmonton Symptom Assessment- revised scale (ESAS-R), a 10-item measure to assess symptoms. The ESAS-R score range 0-100 with higher scores indicating worse symptom burden.
Change in Symptom Management | Baseline to 3 months
  Assessed by PROMIS - Self Efficacy for Managing Symptoms, a 4-item set of person-centered measures that evaluates and monitors physical health.
Change in Hope | Baseline to 3 months
  Assessed by the Herth Hope Index (HHI), which measures various dimensions of hope using a 4-point Likert scale that ranges from 1 (strongly disagree) to 4 (strongly agree) with items #3 and #6 reverse-coded.
Change in Coping | Baseline to 3 months
  Assessed by Brief Cope, a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event.
Change in Social Isolation | Baseline to 3 months
  Assessed by PROMIS - Social Isolation, a 4-item set of person-centered measures that evaluates and monitors social wellbeing.
Change in Financial Well-Being | Baseline to 3 months
  Assessed by Comprehensive Score for Financial Toxicity (COST), an 11-item instrument measures financial toxicity.
Change in Anxiety | Baseline to 3 months
  Assessed by Patient Health Questionnaire-4 (PHQ-4), a brief self-report validated questionnaire that consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2).
Change in Depression | Baseline to 3 months
  Assessed by Patient Health Questionnaire-4 (PHQ-4), a brief self-report validated questionnaire that consists of a 2-item depression scale (PHQ-2) and a 2-item anxiety scale (GAD-2).
Change in Prognostic Awareness | Baseline to 3 months
  Assessed by Prognostic Awareness Impact Scale (PAIS), a 34-item instrument measuring prognostic awareness and its psychological and behavioral impact.
Change in Spiritual Wellbeing | Baseline to 3 months
  Assessed by Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12 Item Scale (FACIT - Sp), a 12-item questionnaire that measures spiritual well-being in cancer and other chronic illnesses.
Change in Perception of the Nurse-Patient Relationship | At 3 months
  Assessed by the RELATE scale, a 17-item instrument that measures patient perceptions of the nurse-patient relationship.
Survival | Through study completion, an average of two years
  Calculated by log rank test, cox proportional hazard modeling, and Kaplan Meyer plots.
Number of Days on Trial | Through study completion, an average of two years
  Calculated by log rank test, cox proportional hazard modeling, and Kaplan Meyer plots.
Percentage of Participants Completing Dose-Limiting Toxicity (DLT) Period | 1 year
Number of Emergency Department Visits | Through study completion, an average of two years
Utilization of Supportive Care Services | Through study completion, an average of two years
  Calculated by log rank test, cox proportional hazard modeling, and Kaplan Meyer plots.
Percentage of Hospice Utilization | Through study completion, an average of two years

CONTACTS AND LOCATIONS:
Overall Officials: Debra Lundquist, PhD, RN, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Debra Lundquist, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation